CLINICAL TRIAL: NCT00348114
Title: Transplantation of Ex-Vivo Expanded Human Limbal Epithelial Stem Cells (LSC) on Amniotic Membrane (AM) for Limbal Stem Cell Deficiency (LSCD).
Brief Title: Transplantation of Cultivated Limbal Epithelium on Amniotic Membrane for Limbal Stem Cell Deficiency
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R260/05/2002
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2002-01

CONDITIONS: Ocular Surface Disease
Keywords: autologous; transplantation ex-vivo expanded limbal epithelium; limbal deficiency

INTERVENTIONS:
Procedure: Transplantation of cultivated limbal epithelium

SUMMARY:
To evaluate the effectiveness of autologous (tissue from fellow eye) transplantation of cultivated limbal epithelium on amniotic membrane to treat severe surface irregularity and scarring of the corneal surface.

DETAILED DESCRIPTION:
The corneal epithelium is under constant cell-turnover,and it has been shown that the limbus is the ultimate source of epithelial renewal. Significant damage to limbal cells causes a disease state called limbal stem cell deficiency(LSCD),characterized by different extents of conjunctival overgrowth onto cornea, vascularization, chronic inflammation, and poor epithelial integrity.

In unilateral LSCD, the damaged corneal surface may be reconstructed using two large segments of healthy limbal tissue (of approximately 6-8mm by 1mm) from the fellow eye in the procedure of conventional limbal transplantation.This may however compromise ocular surface integrity of the healthy eye depending on the amount of donated limbus. In more recent years, it has been possible to "save" limbal tissue by obtaining only a very small limbal biopsy (2mm by 1mm) from the fellow healthy eye which is "expanded" into a viable sheet of limbal cells via laboratory cultivation.This cultivated sheet of cells is transplanted to treat the damaged ocular surface.

This study is a prospective nonrandomized trial which evaluates the efficacy of transplantation of autologous ex-vivo expanded limbal epithelium on intact amniotic membrane for unilateral total limbal stem cell deficiency.

ELIGIBILITY:
Inclusion Criteria:

* unilateral total limbal stem cell deficiency with normal fellow eye, or minimally damaged fellow eye (less than 1/3 limbus affected)

Exclusion Criteria:

* systemic disease affecting both eyes such as Stevens-Johnson syndrome

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8
Dates: Start 2002-05; Study Completion 2006-05

PRIMARY OUTCOMES:
Snellen visual acuity
corneal epithelial integrity and stability

SECONDARY OUTCOMES:
extent of retarding recurrent neovascularisation

CONTACTS AND LOCATIONS:
Overall Officials: Seng-Ei Ti, FRCS(Ed), Principal Investigator — Singapore National Eye Centre; Donald TH Tan, FRCS(G), Study Director — Singapore Eye Research Institute and Singapore National Eye Centre

REFERENCES:
- [Background] Ti SE, Anderson D, Touhami A, Kim C, Tseng SC. Factors affecting outcome following transplantation of ex vivo expanded limbal epithelium on amniotic membrane for total limbal deficiency in rabbits. Invest Ophthalmol Vis Sci. 2002 Aug;43(8):2584-92. PMID 12147589
- [Background] Tsai RJ, Li LM, Chen JK. Reconstruction of damaged corneas by transplantation of autologous limbal epithelial cells. N Engl J Med. 2000 Jul 13;343(2):86-93. doi: 10.1056/NEJM200007133430202. PMID 10891515